CLINICAL TRIAL: NCT04257240
Title: Does Vascular Occlusion in Liver Resections Predispose to Recurrence of Malignancy in the Liver Remnant Due to Ischemia/Reperfusion Injury?
Brief Title: Recurrence of Liver Malignancy After Ischemia/Reperfusion Injury
Acronym: annie-liver
Status: Completed | Type: Observational
Sponsor: Aretaieion University Hospital (Other)
Responsible Party: Principal Investigator, Dr Kassiani Theodoraki, Associate Professor of Anesthesiology, Aretaieion University Hospital
Other Study IDs: liver IR
Record Dates: First submitted 2020-02-02; First posted 2020-02-05 (Actual); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Ischemic Reperfusion Injury; Liver Injury; Cancer Recurrence; Malignancy; Liver Cancer
Keywords: ischemia reperfusion injury; liver surgery; cancer recurrence; malignancy; hepatectomy
MeSH Terms: conditions — Neoplasms; Liver Neoplasms; Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- study group: patients subjected to major hepatectomy with vascular control of blood inflow and outflow of the whole liver
  Interventions: Procedure: selective hepatic vascular exclusion
- control group: patients subjected to major hepatectomy by selectively clamping the portal and hepatic vessels only of the lobe harboring the tumor
  Interventions: Procedure: semielective hepatic vascular exclusion

INTERVENTIONS:
Procedure: selective hepatic vascular exclusion — major hepatectomy with vascular control of blood inflow and outflow of the whole liver
  Groups: study group
Procedure: semielective hepatic vascular exclusion — major liver resection by selectively clamping the portal and hepatic vessels only of the lobe harboring the tumor
  Groups: control group

SUMMARY:
Severe ischemic changes of the liver remnant after hepatectomy could expedite tumor recurrence on the residual liver. Our study aimed at assessing the effect of warm ischemic/reperfusion (I/R) injuries on surgery-to-local recurrence interval and patient overall survival, during major hepatectomies under inflow and outflow vascular control.

DETAILED DESCRIPTION:
One hundred and eighteen patients were subjected to liver resection under total inflow and outflow vascular clamping and were assigned as study group. These individuals were retrospectively matched to 112 counterparts, who underwent liver surgery applying inflow and outflow vascular clamping only of the segment harboring the tumor, sparing the liver remnant from any I/R injury (control group). The two cohorts were compared regarding recurrence-free survival and overall survival.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* American Society of Anesthesiologists (ASA) distribution I to III
* Patients scheduled for major liver resection (≥3 segments)

Exclusion Criteria:

* patients with extrahepatic disease
* patients with metastatic liver tumors

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: retrospective analysis of an internal hepatectomy database
Sampling Method: Non-Probability Sample
Enrollment: 230 (Actual)
Dates: Start 2000-01-01 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2012-12-31 (Actual)

PRIMARY OUTCOMES:
time to malignant recurrence | from time of operation until time of malignant recurrence, assessed up to 15 years
  recurrence-free survival
time to death | from time of operation until time of death, assessed up to 20 years
  overall survival

SECONDARY OUTCOMES:
aspartate aminotrasferase (AST) levels | second postoperative day
  aspartate aminotransferase levels

CONTACTS AND LOCATIONS:
Overall Officials: Kassiani Theodoraki, PhD, Principal Investigator — Aretaieion University Hospital

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Smyrniotis V, Farantos C, Kostopanagiotou G, Arkadopoulos N. Vascular control during hepatectomy: review of methods and results. World J Surg. 2005 Nov;29(11):1384-96. doi: 10.1007/s00268-005-0025-x. PMID 16222453
- [Background] Smyrniotis VE, Kostopanagiotou GG, Contis JC, Farantos CI, Voros DC, Kannas DC, Koskinas JS. Selective hepatic vascular exclusion versus Pringle maneuver in major liver resections: prospective study. World J Surg. 2003 Jul;27(7):765-9. doi: 10.1007/s00268-003-6978-8. PMID 14509502
- [Background] Huang J, Tang W, Hernandez-Alejandro R, Bertens KA, Wu H, Liao M, Li J, Zeng Y. Intermittent hepatic inflow occlusion during partial hepatectomy for hepatocellular carcinoma does not shorten overall survival or increase the likelihood of tumor recurrence. Medicine (Baltimore). 2014 Dec;93(28):e288. doi: 10.1097/MD.0000000000000288. PMID 25526466
- [Background] Liu L, Ren ZG, Shen Y, Zhu XD, Zhang W, Xiong W, Qin Y, Tang ZY. Influence of hepatic artery occlusion on tumor growth and metastatic potential in a human orthotopic hepatoma nude mouse model: relevance of epithelial-mesenchymal transition. Cancer Sci. 2010 Jan;101(1):120-8. doi: 10.1111/j.1349-7006.2009.01363.x. Epub 2009 Sep 14. PMID 19832842
- [Background] Serracino-Inglott F, Habib NA, Mathie RT. Hepatic ischemia-reperfusion injury. Am J Surg. 2001 Feb;181(2):160-6. doi: 10.1016/s0002-9610(00)00573-0. PMID 11425059
- [Background] Man K, Ng KT, Lo CM, Ho JW, Sun BS, Sun CK, Lee TK, Poon RT, Fan ST. Ischemia-reperfusion of small liver remnant promotes liver tumor growth and metastases--activation of cell invasion and migration pathways. Liver Transpl. 2007 Dec;13(12):1669-77. doi: 10.1002/lt.21193. PMID 18044786
- [Background] Ozaki M, Todo S. Surgical stress and tumor behavior: impact of ischemia-reperfusion and hepatic resection on tumor progression. Liver Transpl. 2007 Dec;13(12):1623-6. doi: 10.1002/lt.21230. No abstract available. PMID 18044752
- [Background] Cho JY, Han HS, Choi Y, Yoon YS, Kim S, Choi JK, Jang JS, Kwon SU, Kim H. Association of Remnant Liver Ischemia With Early Recurrence and Poor Survival After Liver Resection in Patients With Hepatocellular Carcinoma. JAMA Surg. 2017 Apr 1;152(4):386-392. doi: 10.1001/jamasurg.2016.5040. PMID 28052154
- [Background] Portolani N, Coniglio A, Ghidoni S, Giovanelli M, Benetti A, Tiberio GA, Giulini SM. Early and late recurrence after liver resection for hepatocellular carcinoma: prognostic and therapeutic implications. Ann Surg. 2006 Feb;243(2):229-35. doi: 10.1097/01.sla.0000197706.21803.a1. PMID 16432356
- [Derived] Theodoraki K, Papadoliopoulou M, Petropoulou Z, Theodosopoulos T, Vassiliu P, Polydorou A, Xanthakos P, Fragulidis G, Smyrniotis V, Arkadopoulos N. Does vascular occlusion in liver resections predispose to recurrence of malignancy in the liver remnant due to ischemia/reperfusion injury? A comparative retrospective cohort study. Int J Surg. 2020 Aug;80:68-73. doi: 10.1016/j.ijsu.2020.06.019. Epub 2020 Jun 30. PMID 32619621